CLINICAL TRIAL: NCT03440203
Title: Prevalence of Peripheral Neuropathy and Its Impact on Activities of Daily Living in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Mi Mi Thet Mon Win, Graduate Student, Okayama University
Other Study IDs: D16-05; Ethics/DMR/2017/049 (Other: Department of Medical Research, Myanmar)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Neuropathy Peripheral; Activities of Daily Living

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- no Diabetic neuropathy
  Interventions: Other: difficult activities of daily living in each group
- Diabetic peripheral neuropathy
  Interventions: Other: difficult activities of daily living in each group
- Diabetic peripheral neuropathic pain
  Interventions: Other: difficult activities of daily living in each group

INTERVENTIONS:
Other: difficult activities of daily living in each group — Compare the severity of pain by the severity of diabetic peripheral neuropathy. Compare the difficulties in ADLs in three group of diabetic patients
  Other Names: severity of pain in each group

SUMMARY:
The trend of diabetes prevalence was increased by comparing these two national surveys in 2009 and 2014. However, the studies only focused on the prevalence and risk of diabetes and non-communicable diseases in Myanmar. The study focused on the common complications of Diabetic Peripheral Neuropathy (DPN) is rare. The studies in other countries showed high prevalence rate and under-diagnosis of DPN. Most of the patients with DPN did not complain about their symptoms because of without prominent symptoms. DPN is the major complication of diabetes. According to the international studies, DPN has the hidden epidemic and is the common causes which can lead to disability and decreased the quality of life in diabetes. Therefore, the study focused on the prevalence of DPN and its impact on the ADLs is obligatory as the descriptive study to explore the actual situation.

Nursing care is not only for the patients in the hospital but also for the people in the community. Moreover, the nurses have to focus on all levels of prevention. Diabetes is the lifelong diseases and accessibility of health care for everyone with diabetes is a very important issue in the era with increased prevalence of diabetes. Therefore, we all have to focus not only on the primary prevention but also on the secondary and tertiary prevention of diabetes. The secondary and tertiary prevention in the diabetic patients also means the primary prevention of other diseases and disabilities (the complications of diabetes). For diabetic neuropathic patients, maintaining normal daily living is very important liked everyone.

The objective of this study is to evaluate the prevalence of DPN and DPNP in type 2 diabetic patients and impact on the activities of daily living. The descriptive, cross-sectional study design will be used in this study. The inclusion criteria are the person aged over 25 years of age who had already diagnosed type 2 diabetes mellitus, taking any anti-glycemic treatment. The persons who are suffering from neuropathy and neuropathic pain other than diabetes, severe illness of diabetic patients, mental illness and alcoholism will be excluded from this study. The patients who meet the inclusion criteria and come to outpatient diabetic clinics at YGH, NOGH, EYGH, and WYGH will be chosen as a sample after obtaining informed consent.

Data collection will be done at this outpatients diabetic clinic of these four hospitals. This study has already obtained ethical clearance from Nursing Science Ethical Review Committee, Graduate School of Health Sciences, Okayama University, Japan with the review number D1605. It will be carrying out after obtaining approval from Department of Medical Research, Myanmar. At the outset, informed consent will be obtained with detailed information about the purpose of research, the part they need to participate, possible benefits and their rights to withdraw.

ELIGIBILITY:
Inclusion Criteria:

* people aged over 25 years of age who have already been diagnosed with type 2 diabetes mellitus, and who are taking anti-glycemic treatment

Exclusion Criteria:

* people who are suffering from neuropathy and neuropathic pain other than diabetes, severe illness of diabetic patients, mental illness and alcoholism

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients went to the diabetic clinic at the outpatient department of Yangon General Hospital (YGH), North-Okkalapa General Hospital (NOGH), East Yangon General Hospital (EYGH), and West Yangon General Hospital (WYGH) in Myanmar used as the sample. These four hospitals are providing outpatient services for diabetics on selected weekdays. Most of the patients who are receiving the care are from Yangon Region.
Sampling Method: Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-10-22 (Actual)

PRIMARY OUTCOMES:
Activities of daily living | on the days of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Mi Mi Thet Mon Win, PhD student, Principal Investigator — Graduate School of Health Sciences, Okayama University
Locations (1):
- Okayama University, Okayama, Japan